CLINICAL TRIAL: NCT01200069
Title: Intravenous Ibuprofen/Caldolor for Post-Electroconvulsive Therapy Myalgia
Brief Title: IV Ibuprofen for Post-Electroconvulsive Therapy Myalgia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: unable to increase to target enrollment
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0120100189
Record Dates: First submitted 2010-08-19; First posted 2010-09-13 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2017-03-29 (Actual); Status verified 2015-03

CONDITIONS: Depression, Myalgia
Keywords: depression,myalgia
MeSH Terms: conditions — Depression; Myalgia | interventions — Ringer's Lactate; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sugar water (Placebo Comparator): 500 milliliters of intravenous ringers lactate administered over 30 minutes prior to ECT for treatments 1,2 and 3
  Interventions: Drug: Placebo infusion
- Ibuprofen (Active Comparator): 300mg/8milliliters of intravenous ibuprofen/caldolor over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments # 1, 2 and 3
  Interventions: Drug: ibuprofen intravenous

INTERVENTIONS:
Drug: Placebo infusion — Identically appearing placebo dose administered IV prior to ECT and subsequently on ECT treatments 2 and 3
  Other Names: lactated ringers
  Arms: Sugar water
Drug: ibuprofen intravenous — IV ibuprofen 800mg/8ml given over 30 minutes prior to ECT and subsequently on ECT treatments 2 and 3
  Other Names: Caldolor
  Arms: Ibuprofen

SUMMARY:
Post-procedure myalgia (muscle ache) is a well-known and common complication of Electro-convulsive Treatment (ECT). Myalgias are a serious concern of patients and occur in approximately 50% of these cases. The pain is usually described as muscle soreness, similar to that resulting from strenuous exercise. The myalgias typically begin shortly after the procedure, lasting approximately 2-7 days in total. A recent study reported that 89% of patients considered prevention significant and would be willing to pay a median of $33 out of pocket to avoid this side effect. In addition to patient discomfort, myalgias can have a further financial burden if these patients are unable to return to work or resume previous daily activities in the days following the procedure. An agent that could treat and possibly even prevent these myalgias has the potential to be very beneficial to these patients. IV ibuprofen (trade name Caldolor) is a novel therapeutic modality approved by the US Food and Drug Administration (FDA) in June 2009 for the treatment of mild to moderate pain, as an adjunct to opioid analgesics, and for the reduction of fever.

DETAILED DESCRIPTION:
IV ibuprofen (trade name Caldolor) is a novel therapeutic modality approved by the US Food and Drug Administration (FDA) in June 2009 for the treatment of mild to moderate pain, as an adjunct to opioid analgesics, and for the reduction of fever. Ibuprofen is a non-steroidal anti-inflammatory drug (NSAID), which produces its effect through inhibition of the enzyme cyclooxygenase (COX). There are at least 2 variations of cyclooxygenase (COX-1 and COX-2) and ibuprofen non-selectively inhibits both, thus decreasing prostaglandin synthesis. This action gives ibuprofen its analgesic, anti-pyretic, and anti-inflammatory properties. NSAIDs have an established history of efficacy in the treatment of both acute and chronic somatic pain. Caldolor, being an intravenous formulation, offers a distinct advantage in patients who either are unable to take medications orally or are fasting preoperatively.

Post-procedure myalgia is a well-known and common complication of ECT. Although the exact etiology is unknown, the myalgias are believed to result from a combination of succinylcholine administration and the seizure activity induced by the ECT procedure itself. Succinylcholine-induced postoperative myalgias are a well-known phenomenon, initially described in the early 1950's. The exact pathogenesis is unknown, with muscle damage from succinylcholine-induced fasciculations or calcium-mediated phospholipase A2 activation and prostaglandin production being proposed as possible etiologies. The latter mechanism provides the rationale for using NSAID therapy. However, succinylcholine is unlikely to be the only factor involved in the development of myalgias following ECT, as a recent study showed that dose adjustments to succinylcholine did not affect rates of myalgia in these patients. Furthermore, seizures can also cause direct muscle injury and there have been reports of muscle pain after ECT both with and without succinylcholine.

A thorough literature search using Medline, Ovid, and scholar.google failed to find any research articles evaluating pretreatment therapy for myalgias in post-ECT patients. The current practice for the treatment of myalgias following ECT has been extrapolated from research on succinylcholine-induced myalgia in post-surgical patients. Previous studies have shown at least partial efficacy with pretreatment of nondepolarizing neuromuscular blocking agents, benzodiazepines, sodium channel blockers (predominantly lidocaine), and nonsteroidal anti-inflammatory drugs. The nature of the ECT procedure itself makes several of these modalities undesirable. Both Lidocaine and benzodiazepines can alter the seizure threshold and the short duration of the procedure possibly increases the risks associated with longer acting nondepolarizing muscle relaxants (ie. blurred vision, diplopia, difficulty breathing and swallowing). Therefore, the options for pretreatment are limited. In addition, a recent meta-analysis of randomized trials determined NSAIDs to cumulatively have the best efficacy of any pretreatment therapy in the prevention of post-procedural myalgias. Due to its intravenous formulation, some practitioners have administered ketorolac to ECT patients before the procedure. However, despite a proven efficacy in myalgia prevention shown by NSAIDs as a class, a study specifically examining the use of ketorolac in this regard failed to show any benefit. The use of Ibuprofen has yet to be examined.

Myalgias are a serious concern of patients and occur in approximately 50% of these cases. The pain is usually described as muscle soreness, similar to that resulting from strenuous exercise. The myalgias typically begin shortly after the procedure, lasting approximately 2-7 days in total. A recent study reported that 89% of patients considered prevention significant and would be willing to pay a median of $33 out of pocket to avoid this side effect. In addition to patient discomfort, myalgias can have a further financial burden if these patients are unable to return to work or resume previous daily activities in the days following the procedure. An agent that could treat and possibly even prevent these myalgias has the potential to be very beneficial to these patients.

Experimental Plan:

The study will be a prospective, randomized, double-blinded placebo-controlled clinical trial. The subject population will consist of patients undergoing first time electroconvulsive therapy, ranging in age from 18 to 80 years. Subjects will be given a Mini-Mental State Examination at the time of their presentation for ECT to assess their cognitive ability. If the patient consents and fits the inclusion criteria, patients will be randomized to one treatment modality, which they will receive for the first three treatment sessions. The subject and the person collecting the data will both be blinded as to what treatment modality the subject belongs to. The patients will be divided into two groups, Group 1 and Group 2. Group 1 will be treated with IV ibuprofen 800mg/8ml given over 30 minutes, prior to induction for ECT; while Group 2 will receive an identically appearing placebo dose, also administered IV, over that same time period. Both groups will receive a standardized anesthetic consisting of methohexital at 1 mg/kg IV for induction and succinylcholine 1 mg/kg IV for muscle paralysis. Other medications (eg. anticholinergic or antihypertensive drugs) will be administered at the discretion of the anesthesiologist. ECT will be administered by the psychiatrist in order to achieve a seizure with a motor component of > 15 second duration. Patients will be transported to the recovery room for post-anesthesia care. Rescue analgesics (Tylenol 500mg PO, Tylenol with codeine 300/30mg PO, Fentanyl 25 mcg IV) will be available to any patient with complaints of myalgia or headache pain of VAS >4.

Measurement Tools:

Severity of myalgias will be assessed based on a self-reported assessment utilizing a numerical rating scale (NRS). The scale will be rated as 0 meaning no pain at all and 10 meaning that pain is so severe as to interfere with daily activities.

Questionnaire:

Do you have any muscle aches or pain right now? If yes, how would you rate that muscle ache/pain on a scale of 0 to 10, with 0 being no pain and 10 being pain that is the worst imaginable?

Example:

0 = No pain 1-3 = Mild Pain (nagging, annoying, little interference with everyday activities) 4-6 = Moderate Pain (interferes significantly with everyday activities) 7-10 = Severe Pain (unable to perform everyday activities) Have you had to take any medications to treat your muscle aches? If yes, what medication did you take? How many pills? What was the strength of the medication? Do you have a headache right now? If yes, how would you rate that headache on a scale of 0 to 10, with 0 being no pain and 10 being pain that is the worst imaginable?

Measurements:

Each patient will have a self-reported numerical pain score assessed at baseline before therapy, 1 hour post-ECT, 6 hours post-ECT, 24 hours post-ECT, and finally at 48 hours post-ECT. The 6, 24 and 48 hour post-ECT assessments will be conducted via a telephone conversation. The use of rescue analgesics during recovery will also be documented as well as time from the end of procedure to discharge. The presence of headache will also be documented in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing informed consent
* American Society Anesthesiologists (ASA) rating I-III
* Subjects age 18-80 capable of providing consent.
* Subjects undergoing electroconvulsive therapy using succinylcholine as the sole neuromuscular blocking agent.
* Subjects who have scored ≥23 on the Mini-Mental State Examination.

Exclusion Criteria:

* Subjects who have had a recent thrombotic event, myocardial infarction or stroke or episode of Congestive Heart Failure (CHF) within less than 3 months.
* Subjects who have had a recent cardiovascular surgery within the last 3 months.
* Subjects with active Gastrointestinal bleeding
* Subjects who have asthma, itching or allergic type reaction following aspirin or other NSAID administration
* Subjects with a known hypersensitivity to ibuprofen
* Subjects with heart failure, bleeding disorders or kidney failure
* Subjects taking aspirin, Angiotensin converting enzyme (ACE) inhibitors, or anticoagulants within one month.
* Subjects with any devices used to treat pain (intrathecal pumps, spinal cord stimulators etc)
* Subjects with a history of fibromyalgia or chronic myositis
* Subjects who are pregnant
* Subjects who do not have a phone
* Subjects who have had previous ECT
* Subjects receiving toradol (Ketorolac)
* Subjects with reported renal disease within less than 3 months.
* Subjects who have had previous electroconvulsive therapy within the last 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vasanti Tilak, MD, Principal Investigator — UMDNJ-NJMS
Locations (1):
- University Hospital, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited following assigned schedule date and time for first ECT treatment, Procedure took place in Medical Special procedure unit (same day service)
Groups:
- Sugar Water: 500 mL of ringers lactate over 30 minutes to be administered prior to ECT for treatments 1,2 and 3
  Placebo infusion: Identically appearing placebo dose administered IV prior to ECT and subsequently on ECT treatments 2 and 3
- Ibuprofen: 800mg/8mL of intravenous ibuprofen over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments # 1, 2 and 3
  ibuprofen intravenous: IV ibuprofen 800mg/8ml given over 30 minutes prior to ECT and subsequently on ECT treatments 2 and 3
Period: Overall Study
Arm/Group | Sugar Water | Ibuprofen
Started | 8 | 6
Completed | 8 | 5
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Water | Ibuprofen | Total
Number analyzed (Participants) | 8 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 5 | 13
  >=65 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 8 | 6 | 14
Mini Mental State Examination >23 [Number; unit: participants] — examination of participants to confirm cognitive ability. Questions such as who is the president, what is the day of the week, the date. The scale is from 0-30. Value of 24 or higher indicates absence of cognitive impairment
  participants | 8 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Subject Self Reported Numerical Rating of Incidence and Severity of Post-Electroconvulsive Therapy Myalgias After Treatment 1
Description: subject self reporting rating scale for severity of myalgias utilizing numeric rating scale 0= no pain, 1-3= mild pain, annoyance with little interference with Activities of Daily Living (ADL), 4-6= moderate (interferes significantly with ADL, 7-10 = severe pain unable to perform ADL
Time Frame: Treatment day 1 at 1hour, 6 hour, 24 hours, 48 hours
Population: subjects report at one hour following treatment
Measure: Median (Full Range); unit: units on a scale
Groups:
- Sugar Water-one Hour After Treatment #1: 500 mL of ringers lactate over 30 minutes to be administered prior to ECT for treatment 1, at one hour following procedure
- Ibuprofen One Hour After Treatment #1: 800mg/8mL of intravenous ibuprofen over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments # 1, 2 and 3
  subject report of myalgia one hour after completion of procedure number 1
- Sugar Water 6 Hours After Procedure #1: Subject reported myalgia 6 hours after completion of treatment # 1,
- Ibuprofen 6 Hours After Treatment #1: subject reported myalgia 6 hours after treatment 1
- Sugar Water 24 Hours After Treatment #1: subject reported myalgia 24 hours after completion of procedure 1
- Ibuprofen 24 Hours After Treatment 1: subject reported myalgia 24 hours after procedure 1
- Sugar Water 48 Hours After Procedure 1: subject reported myalgia 48 hours after procedure 1
- Ibuprofen 48 Hours After Treatment 1: subject reported myalgia 48 hours after treatment day 1
Arm/Group | Sugar Water-one Hour After Treatment #1 | Ibuprofen One Hour After Treatment #1 | Sugar Water 6 Hours After Procedure #1 | Ibuprofen 6 Hours After Treatment #1 | Sugar Water 24 Hours After Treatment #1 | Ibuprofen 24 Hours After Treatment 1 | Sugar Water 48 Hours After Procedure 1 | Ibuprofen 48 Hours After Treatment 1
Number analyzed (Participants) | 8 | 6 | 8 | 6 | 8 | 6 | 8 | 6
units on a scale | 2 [0 to 4] | 0 [0 to 0] | 7.5 [5 to 10] | 1.5 [0 to 3] | 2.5 [2 to 5] | .5 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]

2. Primary Outcome: Myalgia Reported on Treatment Day 2
Description: Subject self reported numerical rating of incidence and severity of post ECT Myalgia after treatment day 2 0=no pain, 1-3=mild pain (annoying, little interference with ADL), 4-6= moderate,( interferes significantly with ADL) 7-10 severe pain (unable to perform everyday activities)
Time Frame: 1 hour, 6 hours, 24 hours & 48 hours following procedure
Measure: Median (Full Range); unit: units on a scale
Groups:
- Sugar Water-one Hour After Treatment 2: 500 mL of ringers lactate over 30 minutes to be administered prior to ECT for treatments 2
  Placebo infusion: Identically appearing placebo dose administered IV prior to ECT and subsequently on ECT treatment day 2
- Ibuprofen One Hour After Treatment #2: 800mg/8mL of intravenous ibuprofen over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments # 2 one hour after treatment
  ibuprofen intravenous: IV ibuprofen 800mg/8ml given over 30 minutes prior to ECT treatment day 2
- Sugar Water 6 Hours After Procedure #2; Ibuprofen 6 Hours After Treatment #2: Subject reported myalgia 6 hours after completion of treatment #2
- Sugar Water 24 Hours After Treatment #2; Ibuprofen 24 Hours After Treatment #2: Subject reported myalgia 24 hours after completion of treatment #2
- Sugar Water 48 Hours After Treatment 2; Ibuprofen 48 Hours After Treatment 2: Subject reported myalgia 48 hours after completion of treatment #2
Arm/Group | Sugar Water-one Hour After Treatment 2 | Ibuprofen One Hour After Treatment #2 | Sugar Water 6 Hours After Procedure #2 | Ibuprofen 6 Hours After Treatment #2 | Sugar Water 24 Hours After Treatment #2 | Ibuprofen 24 Hours After Treatment #2 | Sugar Water 48 Hours After Treatment 2 | Ibuprofen 48 Hours After Treatment 2
Number analyzed (Participants) | 8 | 5 | 8 | 5 | 8 | 5 | 8 | 5
units on a scale | 1.5 [0 to 3] | 0 [0 to 0] | 0 [0 to 0] | 1.5 [0 to 3] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

3. Primary Outcome: Myalgia Reported After Treatment #3
Description: Subject self reported severity of myalgia based on a self reported assessment utilizing numeric rating scale 0=no myalgia, 1-3=mild myalgia (annoying, little interference with ADL);4-6=moderate (interferes significantly with ADL); 7-10 severe myalgia(unable to perform every day activities)
Time Frame: 1 hour, 6 hour, 24 hour, 48 hour after 3rd ECT treatment
Measure: Median (Full Range); unit: units on a scale
Groups:
- Sugar Water-one Hour After Treatment 3: 500 mL of ringers lactate over 30 minutes to be administered prior to ECT for treatments 3
  Placebo infusion: Identically appearing placebo dose administered IV prior to ECT and subsequently on ECT treatment day 2
- Ibuprofen One Hour After Treatment #3: 800mg/8mL of intravenous ibuprofen over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments # 3 one hour after treatment
  ibuprofen intravenous: IV ibuprofen 800mg/8ml given over 30 minutes prior to ECT treatment day 2
- Sugar Water 6 Hours After Procedure #3; Ibuprofen 6 Hours After Treatment #3: Subject reported myalgia 6 hours after completion of treatment #3
- Sugar Water 24 Hours After Treatment #3; Ibuprofen 24 Hours After Treatment #3: Subject reported myalgia 24 hours after completion of treatment #3
- Sugar Water 48 Hours After Treatment 3; Ibuprofen 48 Hours After Treatment 3: Subject reported myalgia 48 hours after completion of treatment #3
Arm/Group | Sugar Water-one Hour After Treatment 3 | Ibuprofen One Hour After Treatment #3 | Sugar Water 6 Hours After Procedure #3 | Ibuprofen 6 Hours After Treatment #3 | Sugar Water 24 Hours After Treatment #3 | Ibuprofen 24 Hours After Treatment #3 | Sugar Water 48 Hours After Treatment 3 | Ibuprofen 48 Hours After Treatment 3
Number analyzed (Participants) | 8 | 5 | 8 | 5 | 8 | 5 | 8 | 7
units on a scale | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Subject Self Reported Numerical Rating of Incidence and Severity of Post Electroconvulsive Therapy Headache After Treatment Day 1
Description: Subject self reported numerical rating of incidence and severity of Post ECT pain score for headache at 1, 6, 24 and 48 hours post procedure. Pain Rating 0= no pain, 2-4=moderate pain, 5-7=distressing severe pain, 8-9=intense very severe pain, 10=unbearable pain
Time Frame: 1 hour, 6 hours, 24 hours & 48 hours following procedure
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Pain Score Sugar Water-one Hour After Treatment 1: 500 mL of ringers lactate over 30 minutes to be administered prior to ECT for treatments 1
  Placebo infusion: Identically appearing placebo dose administered IV prior to ECT and subsequently on ECT treatment day 1
- Pain Score Ibuprofen One Hour After Treatment #1: 800mg/8mL of intravenous ibuprofen over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments # 1 one hour after treatment
  ibuprofen intravenous: IV ibuprofen 800mg/8ml given over 30 minutes prior to ECT treatment day 2
- Pain Score After Sugar Water 6 Hours After Treatment #1; Pain Score Ibuprofen 6 Hours After Treatment #1: Subject reported headache 6 hours after completion of treatment #1
- Pain Score Sugar Water 24 Hours After Treatment #1: Subject reported headache 24 hours after completion of treatment #1
- Pain Score Ibuprofen 24 Hours After Treatment #1: Subjects reported headache 24 hours after completion of treatment #1
- Pain Score Sugar Water 48 Hours After Treatment 1; Pain Score Ibuprofen 48 Hours After Treatment 1: Subjects reported headache 48 hours after completion of treatment #1
Arm/Group | Pain Score Sugar Water-one Hour After Treatment 1 | Pain Score Ibuprofen One Hour After Treatment #1 | Pain Score After Sugar Water 6 Hours After Treatment #1 | Pain Score Ibuprofen 6 Hours After Treatment #1 | Pain Score Sugar Water 24 Hours After Treatment #1 | Pain Score Ibuprofen 24 Hours After Treatment #1 | Pain Score Sugar Water 48 Hours After Treatment 1 | Pain Score Ibuprofen 48 Hours After Treatment 1
Number analyzed (Participants) | 8 | 6 | 8 | 6 | 8 | 6 | 8 | 6
units on a scale | 2.6 [0 to 6] | 1.5 [0 to 5] | 3.1 [3 to 10] | 1.3 [0 to 4] | 3.6 [0 to 5] | .16 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]

5. Secondary Outcome: Incidence and Severity of Headache After ECT Treatment 2
Description: Subject self reported numerical rating of incidence and severity of post ECT headache 0=no pain, 2-4=moderate pain, 5-7= distressing severe pain, 8-9= very severe pain, 10=unbearable pain.
Time Frame: 1 hour, 6 hour, 24 hour and 48 hours
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Ibuprofen One Hour After Treatment #2: 800mg/8mL of intravenous ibuprofen over 30 min in 500mL of ringers lactate to be administered prior to ECT for treatments #2 one hour after treatment
  ibuprofen intravenous: IV ibuprofen 800mg/8ml given over 30 minutes prior to ECT treatment day 2
- Sugar Water 6 Hours After Procedure #2; Ibuprofen 6 Hours After Treatment #2: Subject reported headache 6 hours after completion of treatment #2
- Sugar Water 24 Hours After Treatment #2; Ibuprofen 24 Hours After Treatment #2: Subject reported headache 24 hours after completion of treatment #2
- Sugar Water 48 Hours After Treatment #2; Ibuprofen 48 Hours After Treatment #2: Subject reported headache 48 hours after completion of treatment #2
Arm/Group | Sugar Water-one Hour After Treatment 2 | Ibuprofen One Hour After Treatment #2 | Sugar Water 6 Hours After Procedure #2 | Ibuprofen 6 Hours After Treatment #2 | Sugar Water 24 Hours After Treatment #2 | Ibuprofen 24 Hours After Treatment #2 | Sugar Water 48 Hours After Treatment #2 | Ibuprofen 48 Hours After Treatment #2
Number analyzed (Participants) | 8 | 5 | 8 | 5 | 8 | 8 | 7 | 8
units on a scale | 1.4 [0 to 5] | 1.1 [0 to 4] | 1.55 [0 to 5] | 1 [0 to 5] | .18 [0 to 2] | .14 [0 to 1] | 0 [0 to 0] | .14 [0 to 1]

6. Secondary Outcome: Incidence of Headache & Severity Headache After ECT Treatment #3
Description: Subject self reported numerical rating of incidence and severity of post ECT headache after treatment #3, 0=no pain, 2-4=moderate pain, 5-7=distressing severe pain, 8-9 very serious pain, 10=unbearable pain.
Time Frame: 1 hour after treatment, 6 hours, 24 hours and 48 hours
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Sugar Water 6 Hours After Procedure #3; Ibuprofen 6 Hours After Treatment #3: Subject reported headache 6 hours after completion of treatment #3
- Sugar Water 24 Hours After Treatment #3; Ibuprofen 24 Hours After Treatment #3: Subject reported headache 24 hours after completion of treatment #3
- Sugar Water 48 Hours After Treatment 3; Ibuprofen 48 Hours After Treatment 3: Subject reported headache 48 hours after completion of treatment #3
Arm/Group | Sugar Water-one Hour After Treatment 3 | Ibuprofen One Hour After Treatment #3 | Sugar Water 6 Hours After Procedure #3 | Ibuprofen 6 Hours After Treatment #3 | Sugar Water 24 Hours After Treatment #3 | Ibuprofen 24 Hours After Treatment #3 | Sugar Water 48 Hours After Treatment 3 | Ibuprofen 48 Hours After Treatment 3
Number analyzed (Participants) | 8 | 5 | 8 | 5 | 8 | 5 | 8 | 5
units on a scale | 0 [0 to 0] | .64 [0 to 4] | .28 [0 to 2] | 1 [0 to 6] | 0 [0 to 0] | .16 [0 to 1] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 0-72 hours after each of the 3 treatments
Description: treatment day 1 at 1 hour post ECT procedure subject experienced dizziness
  treatment day 3 at 6 hour post procedure subject reported dizziness
Arm/Group | Sugar Water | Ibuprofen
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/6
Other Adverse Events (participants affected / at risk) | 2/8 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sugar Water (N=8) | Ibuprofen (N=6)
dizzyness (Nervous system disorders) | 2 | 0
vomiting (Gastrointestinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes